CLINICAL TRIAL: NCT02133339
Title: A Phase I, Randomized, Double-blind, Placebo Controlled, Single Ascending Dose Study to Evaluate the Safety and Tolerability of Nebulized, TRN-157 Inhalation Solution in Healthy Subjects
Brief Title: Single Ascending Dose Study of TRN-157 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theron Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRN-157-101
Record Dates: First submitted 2014-05-05; First posted 2014-05-08 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- TRN-157 (Experimental)
  Interventions: Drug: TRN-157
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRN-157
  Arms: TRN-157
Drug: Placebo
  Arms: Placebo

SUMMARY:
This single ascending dose study is to determine and evaluate the safety and tolerability of TRN-157 in approximately 40 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent
2. The subject is male or female 18 to 65 years of age
3. If the subject or subject's partner is of childbearing potential, a medically acceptable form of contraception will be
4. Non-smoker
5. Good general health
6. Willing to abstain from alcohol, caffeine, and xanthine-containing beverages
7. The subject is compliant and available throughout the entire study period

Exclusion Criteria:

1. Current diagnosis, as per subject or investigator or screening assessment, of:

   1. unstable or uncontrolled disease in any organ system (including cardiovascular) on present therapy
   2. history of narrow angle glaucoma
   3. history of alcohol abuse within the past 5 years
   4. history of smoking within the past 6 months
   5. positive result for the alcohol and/or drugs of abuse
   6. weight > 100 kg or < 50 kg
   7. clinically significant abnormal ECG
   8. history of clinically significant (per the Investigator) disease or disorder
   9. any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results
   10. Abnormal vital signs defined as any of the following:

       * Systolic blood pressure ≥ 140 mmHg
       * Diastolic blood pressure ≥ 90mmHg
2. Heart rate < 40 or > 85 beats per minute
3. Fever or other clinically significant physical exam findings
4. Current or history of clinically significant respiratory disease, including asthma, emphysema, chronic bronchitis, or cystic fibrosis
5. History or current symptom(s) of respiratory tract inflammation
6. Inability to perform reproducible spirometry in accordance with American Thoracic Society (ATS) guidelines
7. Abnormal FEV1, FVC, or FEV1/FVC (FEV1 or FVC < 80% of predicted or FEV1/FVC ratio < 0.7)
8. FEV1 variability > 10% between study visits
9. Female of childbearing potential with a positive serum pregnancy test or currently breastfeeding
10. Currently being treated for hypertension or taking any other medications that affect blood pressure significantly
11. Inability to perform acceptable, quality serial spirometry or any other study procedures
12. Positive screen for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, or HIV antibody

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as determined by number of subjects with adverse events | 1 week

SECONDARY OUTCOMES:
Determination of pharmacokinetic parameters | 1 week
  Area Under the Plasma Concentration-Time Curve from Zero to the Time of the Last Measurable Concentration (AUC0-t)
Determination of pharmacokinetic parameters | 1 week
  Area Under the Plasma Concentration-Time Curve from Zero to Infinity (AUC0-inf)
Determination of pharmacokinetic parameters | 1 week
  Peak Plasma Concentration (Cmax)
Determination of pharmacokinetic parameters | 1 week
  Time to Peak Plasma Concentration (tmax)
Determination of pharmacokinetic parameters | 1 week
  Half-Life (t½)
Determination of pharmacokinetic parameters | 1 week
  Elimination Rate Constant (kel)
Determination of pharmacokinetic parameters | 1 week
  Volume of Distribution at Steady State after Non-IV Administration (Vss/F)
Determination of pharmacokinetic parameters | 1 week
  Total Plasma Clearance after Non-IV Administration (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Oren, Study Director — Theron Pharmaceuticals, Inc.
Locations (1):
- Cypress, California, United States